CLINICAL TRIAL: NCT06961838
Title: The Effect of Inspiratory Muscle Training With Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Beyzanur Dikmen, Research Assistant, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ÜsküdarÜ2025
Record Dates: First submitted 2025-04-17; First posted 2025-05-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Substance Abuse Disorder; Exercise; Pulmonary Function; Rehabilitation
Keywords: Substance Use Disorder; Exercise; Rehabilitation; Pulmonary Function; Muscle Training
MeSH Terms: conditions — Substance-Related Disorders; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Experimental): In addition to their standard treatment, individuals in the inspiratory muscle training group will participate in inspiratory muscle training for a total of 30 minutes with a threshold loading device (POWERbreathe®) for 15 minutes twice a day, 5 days a week for 4 weeks under the supervision of a physiotherapist.
  Interventions: Other: Inspiratory muscle training programme
- Control group (Active Comparator): Individuals in the control group will continue their standard treatment.
  Interventions: Other: control group

INTERVENTIONS:
Other: Inspiratory muscle training programme — In addition to their standard treatment, individuals in the inspiratory muscle training group will participate in inspiratory muscle training for a total of 30 minutes with a threshold loading device (POWERbreathe®) for 15 minutes twice a day, 5 days a week for 4 weeks under the supervision of a physiotherapist.
  Arms: Inspiratory muscle training group
Other: control group — Individuals in the control group will continue their standard treatment. No changes will be made in the medical treatments (type, dosage and frequency) of the individuals in both groups (the inspiratory muscle training group and the control group) during the study.
  Arms: Control group

SUMMARY:
The aim was to investigate the effectiveness of inspiratory muscle training on dyspnoea, pulmonary function, respiratory muscle strength, cough capacity, functional exercise capacity, substance craving, depression, anxiety and quality of life in individuals with substance use disorder.

DETAILED DESCRIPTION:
In recent years, substance use has increased among young people in our country, and studies investigating the negative effects of substances on pulmonary health have also increased. It has been emphasized in the literature that the most appropriate features should be determined for the exercise program in the treatment of individuals with SUD. Although studies in the literature have reported that substance use affects respiratory functions and creates a restrictive or obstructive pattern, no study investigating the effects of inspiratory muscle training has been found in the literature. To our knowledge, this study is the first to examine the effects of inspiratory muscle training on respiratory function in individuals with SUD. In our study, it was assumed that inspiratory muscle training could be a simple and inexpensive technique to improve dyspnea, respiratory functions, respiratory muscle strength, cough capacity, and exercise capacity in individuals with SUD, reduce substance cravings, increase quality of life, and reduce depression and anxiety, thus making it suitable for routine clinical use. The aim was to examine the effectiveness of inspiratory muscle training on dyspnea, respiratory functions, respiratory muscle strength, functional exercise capacity, substance craving, anxiety, depression, and quality of life in individuals with substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years

  * Meeting the current Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for Substance Use Disorder
  * Receiving inpatient treatment
  * Substance use for more than one year
  * Being able to follow simple instructions
  * Not having any visual and auditory pathology
  * Being able to cooperate with the devices used.

Exclusion Criteria:

* Failure to comply with the treatment and assessment program
* Participation in a structured physiotherapy/exercise program in the last 6 months
* Presence of current psychotic symptoms
* Presence of any physical disability or medical problem
* Presence of respiratory system problems such as asthma and tuberculosis and infectious health problems (e.g. HIV, hepatitis B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | 4 weeks
  Participants' perceptions of dyspnoea in daily life will be assessed using the Modified Medical Research Council Scale (mMRC), which consists of five statements describing the full range of dyspnoea from none (Grade 0) to almost complete incapacity (Grade 4).
Respiratory Functions (FEV1) | 4 weeks
  Based on ATS and ERS recommendations, a portable spirometer (Cosmed Pony FX, Rome, Italy) will be used to assess pulmonary function testing. At the end of the pulmonary function test, forced expiratory volume in 1 second (FEV1) will be recorded.
Respiratory Functions (FVC) | 4 weeks
  Based on ATS and ERS recommendations, a portable spirometer (Cosmed Pony FX, Rome, Italy) will be used to assess pulmonary function testing. At the end of the pulmonary function test, forced vital capacity (FVC) will be recorded.
Respiratory Functions (FEV1/FVC) | 4 weeks
  Based on ATS and ERS recommendations, a portable spirometer (Cosmed Pony FX, Rome, Italy) will be used to assess pulmonary function testing. At the end of the pulmonary function test, FEV1/FVC ratio will be recorded.
Respiratory Functions (FEF 25-75%) | 4 weeks
  Based on ATS and ERS recommendations, a portable spirometer (Cosmed Pony FX, Rome, Italy) will be used to assess pulmonary function testing. At the end of the pulmonary function test, forced expiratory flow (FEF 25-75%) will be recorded.
Respiratory Functions (PEF) | 4 weeks
  Based on ATS and ERS recommendations, a portable spirometer (Cosmed Pony FX, Rome, Italy) will be used to assess pulmonary function testing. At the end of the pulmonary function test, peak expiratory flow (PEF) will be recorded.
Respiratory Muscle Strength | 4 weeks
  The respiratory muscle strength of the participants will be assessed by maximal inspiratory (MIP) and expiratory intraoral pressures (MEP).
Cough Capacity | 4 weeks
  Participants' peak cough flow will be measured using a Peak Flow Meter (The Mini-Wright Standard, Cartel Business Estate, Edinburgh Way, Harlow) while individuals are making a maximal cough effort after as deep an inspiration as possible.
Functional exercise capacity | 4 weeks
  Functional exercise capacity will be assessed using the 6-Minute Walk Test (6-MWT) performed using standard protocols in accordance with American Thoracic Society guidelines.

SECONDARY OUTCOMES:
Penn Substance Craving Scale | 4 weeks
  It is a 5-item self-report questionnaire developed to assess substance craving over the past week, including frequency, intensity, duration, urgency, and total craving. Each item is rated on a scale of 0 to 6, with a maximum total score of 30 for severe cravings.
Health-related quality of life | 4 weeks
  Health-related quality of life will be assessed with the health-related quality of life Short Form 12 questionnaire. Information from all 12 items is used to calculate the physical component summary and the mental health component summary score. All scores are converted into a standardized score between 0-100. Higher scores indicate better health-related quality of life.
Anxiety and Depression | 4 weeks
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report questionnaire assessing levels of depression (7 items) and anxiety (7 items). Each item is rated on a 4-point Likert scale. Subscale scores were calculated by summing the subscale items (subscale scores range from 0-21), with higher scores indicating greater severity. It has been previously shown that HADS scores equal to or higher than 10 and 7 on the relevant anxiety and depression items, respectively, indicate clinical levels of anxiety and depression in the Turkish population.

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar University, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivasothy P, Brown L, Smith IE, Shneerson JM. Effect of manually assisted cough and mechanical insufflation on cough flow of normal subjects, patients with chronic obstructive pulmonary disease (COPD), and patients with respiratory muscle weakness. Thorax. 2001 Jun;56(6):438-44. doi: 10.1136/thorax.56.6.438. PMID 11359958
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Laszlo G. Standardisation of lung function testing: helpful guidance from the ATS/ERS Task Force. Thorax. 2006 Sep;61(9):744-6. doi: 10.1136/thx.2006.061648. PMID 16936234